CLINICAL TRIAL: NCT03983447
Title: School Intervention to Promote Physical Activity and Reduce the Sedentary Time of Low-income Children Aged 6-13 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pau and Pays de l'Adour (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UPPA (University of Pau)
Record Dates: First submitted 2019-06-03; First posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Physical Activity; Sedentary Behavior; Children; School-based Intervention
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: During the academic year 2016/2017, baseline assessments were carried out in two schools (school A, school B): measures of PA, ST, motors skills, attentional capacity and academic achievement. These assessments were performed in November/December 2016 (First Time - T1) and May/June 2017 (Second time - T2).
  During the academic school year 2017/2018, a school-based intervention to increase PA and reduce ST was realised in School A (measure in November 2017 and May/June 2018). Finally, during the academic school year 2018/2019, a school-based intervention to increase PA and reduce ST was realised in School B (measure only in May/June 2019).
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- School-based intervention to promote Physical Activity (PA) (Experimental): This intervention included :
  1. Physical (Environmental) adaptation of playground
  2. Time adaptation of lunch breaks
  3. Curriculum-based program of children
  4. Workshops and newsletters for parents
  5. Meetings for teachers
  Interventions: Behavioral: School-based intervention to promote PA and reduce ST
- Control (No Intervention): Nothing has changed in the school.

INTERVENTIONS:
Behavioral: School-based intervention to promote PA and reduce ST — This intervention was realized with all the children (1st grade-5th grade) and involved :
  1. Physical (Environmental) adaptation of playgrounds
  2. Time adaptation of lunch breaks
  3. Curriculum-based program for children
  4. Workshops and newsletters for parents
  5. Meetings for teachers
  Arms: School-based intervention to promote Physical Activity (PA)

SUMMARY:
This study is realized in 2 primary schools in the city of Tarbes (France), located in a disadvantaged neighbourhood : 352 children are included in the study.

This study has many goals: 1) to propose an intervention to promote PA (Physical Activity) and reduce ST (Sedentary Time) of children aged 6 to 13 years from a primary school located in a disadvantaged neighbourhood and measures the effectiveness of this intervention (1rst grade-5th grade). This intervention was based on the factors of socio-ecological model related to health behaviours. The levels of PA and ST of the experimental school will be compared to a control school with the realization of pre and post intervention measures. 2) To study the relationships between PA, ST, motors skills, attentional abilities and academic achievement. 3)To realise a descriptive analysis of PA and ST of children in 2nd and 5th grade from France and Spain (observational study). For this goal, an other school in Spain was included in the study (city of Huesca, 60 children).

DETAILED DESCRIPTION:
Physical activity (PA) has decreased drastically in the 21st century in developed and industrialized societies. In 2009, 23.3% of the world's population did not comply with WHO's recommendations for physical activity, reaching real levels of pandemic. Technological advances have contributed to the emergence of new leisure activities, which may preclude the participation in PA and encourage sedentary behaviours. However, it is now well known that PA has numerous benefits on physical, psychological and social health. Thus, promoting PA becomes a necessity for adults and even more for children since healthy habits that are adopted during childhood will last throughout life and predict adult health. Hence, for this last population, 60 minutes of moderate-to-vigorous physical activity (MVPA) per day are recommended in public health guidelines.

A recent project named "Capas-Cité", created in 2012 in Tarbes (France) and in Zaragoza (Spain) realize PA programs and promotion actions that have a beneficial impact on health. These two similar cities have been selected for their geographical proximity and their similarity. These programs are included in research work carried out by the University of Tarbes and the University of Zaragoza that focus on the promotion of PA. "Capas-Cité" project aims to improve the health of disadvantaged population.

The two primary schools (School A and School B) located in the disadvantaged neighbourhood of Tarbes were contacted to participate in the study. Both schools include children from grade 1 (6 years old) to grade 5 (10 years old). They have never benefited from intervention programs on the field of PA and agreed to participate in the project.

During the academic year 2016/2017, baseline assessments were carried out in the two French schools: measures of PA, ST, motors skills, attentional abilities and academic achievement. These assessments were performed in November/December 2016 (First Time - T1) and May/June 2017 (Second time - T2). The measures of attentional abilities involve only children in 2nd, 3th and 4th grade. Children in both schools had to have parental permission to participate in PA, ST and attentional abilities measurements. Motor skills were assessed for all the children at school and their academic achievement were collected.

During the academic school year 2017/2018, School A benefited of an intervention to increase PA and reduce ST. This intervention program involves all the children from grade 1 to grade 5 without parental permission. Families are not required to contribute financially participation in this project. During this intervention year, the same periods of assessment as those carried at baseline were repeated in November/December 2017 (T3) and May/June 2018 (T4). These repeated assessment time provide a first overview of the efficiency of the intervention. The school B has the intervention program during the school year 2018/2019.

Accelerometers were used to measure PA and ST. Accelerometry is a reliable and valid objective to measure PA and ST. Children should wear the accelerometer on the right side of the hip, adjusted with an elastic belt.

In Spain, only observational measures were realised. . A total of 179 children have worn accelerometers for a week. PA and ST were analysed for week end days on one hand and on the other hand according to different periods of time for weekdays: the time before school, lunch, after school and at night.54.97% of the children complied with the MVPA guidelines all days of the week. MVPA represented 67.70±17.83 min.day-1 and ST was 606.14±37.39 min.day-1 for the total sample.

ELIGIBILITY:
Inclusion Criteria:

* Children (girls, boys) aged 5-13 years old

Exclusion Criteria:

* Physical diseases that prevent PA practice

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 350 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Physical Activity (PA) | 7 days
  Units : "counts/minute" and "minutes". Children from grade 1 to 5 who had parental permission to participate in the project carried an accelerometer (Actilife, Pensacola, FL, USA) to assess their usual levels of PA. Accelerometry is a reliable and valid objective to measure PA.
Sedentary Time (ST) | 7 days
  Units : "counts/minute" and "minutes". Children from grade 1 to 5 who had parental permission to participate in the project carried an accelerometer (Actilife, Pensacola, FL, USA) to assess their usual levels of ST. Accelerometry is a reliable and valid objective to measure ST.

SECONDARY OUTCOMES:
Anthropometry: Body Mass Index (BMI) | 10 minutes for each child
  Units : kg/m^2.The weight and height of the children were measured just prior of this test, in each measurement period
Subjective information about family and child | 20 minutes
  Parents participating in the project were asked to complete a questionnaire to obtain some information: age and gender of the child; socioeconomic data measured by the four-item scale "Family Affluence Scale II" (FAS II) (Boyce, Torsheim, Currie et Zambon, 2006). FAS II: 4 item-scale that asks families how many "car/bedrooms/computers" they have and how often they go on holiday. A composite FAS score is calculated for each family summing up the responses to these four items. The sample is then categorised using a three-point ordinal scale where low FAS (score=0,1,2) indicates low affluence, medium FAS (score=3,4,5) indicates medium affluence, and high FAS (score=6,7,8,9) indicates high affluence (Aibar, 2012) ; parental perception of the competence of their children in physical activity practice; sedentary behaviour of the child (time spent playing video games, wa
Standing broad jump (Motor Skills) | 2 hours for each grade
  Units : cm. The test was realized for all children from grade 1 to 5 in a two-hour physical education class. This test of the Eurofit battery measures power and inter-segmental coordination. He stands behind a starting line and jump by throwing his arms forward. Three trials are allowed and only the best performance is analysed.
Plate tapping test (Motor Skills) | 2 hours for each grade
  Units : seconds.The assessment of this test was realized for all children from grade 1 to 5 in a two-hour physical education class. The speed and coordination of the upper limbs is measured. The child is situated in from of a table. Two rubber discs 20 cm in diameter are fixed horizontally on the table, with a gap of 60 cm. A rectangular plate is placed between the two discs. The child puts a hand in the middle of the rectangular plate and touches the discs alternatively as quickly as possible with the other hand, passing over the hand situated in the middle. He performs 25 cycles.
6 x 5m Shuttle Run (Motor Skills) | 2 hours for each grade
  Units: seconds.This test was realized for all children from grade 1 to 5 in a two-hour physical education class.This test was adapted from the 10x5m shuttle test of the Eurofit battery. It measures the speed-coordination of inter-segmental limbs. The specialist evaluates the time needed to cover the distance with a stopwatch.
Cardiorespiratory fitness: 20m shuttle run test | 2 hours for each grade
  Units: seconds.The assessment of motor skills was realized for all children from grade 1 to 5 in a two-hour physical education class.The aerobic capacity of the children was measured with an adapted version of the 20m shuttle run test (Cadenas Sanchez, 2011). The initial speed is reduced at 6.5 km/h and increase according to the laps and the stage numbers.
Academic achievement | 1 hour for each grade
  Units : %. The learning achievement for children from grade 1 to 5 was collected at the beginning of the school year. The percentages of success rate of "reading", "spelling" and "mathematics" were collected.
Attention | 10 minutes for each child
  Units : % and seconds.The computer-based modified Erickson Flanker Task was used (Have et al, 2016). It was designed with the software Superlab 4.5 (AD instruments) by the researcher specialist. This test is a variant version of the classing Flanker-Task (Eriksen et Ericksen, 1974). It permits the measurement of inhibition and cognitive flexibility, which are identified as executive functions and specifically attentional abilities.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aibar A, Bois JE, Generelo E, Zaragoza Casterad J, Paillard T. A cross-cultural study of adolescents' physical activity levels in France and Spain. Eur J Sport Sci. 2013;13(5):551-8. doi: 10.1080/17461391.2012.746733. Epub 2012 Nov 23. PMID 24050473
- [Background] Kriemler S, Meyer U, Martin E, van Sluijs EM, Andersen LB, Martin BW. Effect of school-based interventions on physical activity and fitness in children and adolescents: a review of reviews and systematic update. Br J Sports Med. 2011 Sep;45(11):923-30. doi: 10.1136/bjsports-2011-090186. PMID 21836176
- [Background] Hartmann T, Zahner L, Puhse U, Puder JJ, Kriemler S. Effects of a school-based physical activity program on physical and psychosocial quality of life in elementary school children: a cluster-randomized trial. Pediatr Exerc Sci. 2010 Nov;22(4):511-22. doi: 10.1123/pes.22.4.511. PMID 21242601
- [Background] Rhodes RE, Janssen I, Bredin SSD, Warburton DER, Bauman A. Physical activity: Health impact, prevalence, correlates and interventions. Psychol Health. 2017 Aug;32(8):942-975. doi: 10.1080/08870446.2017.1325486. Epub 2017 May 30. PMID 28554222
- [Background] Scudder MR, Lambourne K, Drollette ES, Herrmann SD, Washburn RA, Donnelly JE, Hillman CH. Aerobic capacity and cognitive control in elementary school-age children. Med Sci Sports Exerc. 2014;46(5):1025-35. doi: 10.1249/MSS.0000000000000199. PMID 24743109
- [Background] Khan NA, Hillman CH. The relation of childhood physical activity and aerobic fitness to brain function and cognition: a review. Pediatr Exerc Sci. 2014 May;26(2):138-46. doi: 10.1123/pes.2013-0125. Epub 2014 Apr 10. PMID 24722921
- [Derived] Bernal CMM, Lhuisset L, Fabre N, Bois J. School-Based Multicomponent Intervention to Promote Physical Activity and Reduce Sedentary Time of Disadvantaged Children Aged 6-10 Years: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Sep 23;9(9):e17815. doi: 10.2196/17815. PMID 32965238